CLINICAL TRIAL: NCT04795024
Title: Effectiveness of Yamamoto's New Skull Acupuncture (YNSA) on Resting State Brain Networks
Brief Title: Effectiveness of YNSA Acupuncture on Brain Networks
Status: Completed | Type: Observational
Sponsor: BDH-Klinik Hessisch Oldendorf (Other)
Responsible Party: Sponsor
Other Study IDs: YNSA-EFF
Record Dates: First submitted 2021-03-09; First posted 2021-03-12 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Acupuncture
Keywords: Resting-state fMRI

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study investigates the effects of a new form of acupuncture (Yamamoto's New Skull Acupuncture [YNSA]) on resting-state brain networks. Therefore, two resting-state fMRI scans are measured (one without and one with acupuncture needles) in healthy adults. It is expected that acupuncture is associated with changes in functional connectivity within different brain networks.

DETAILED DESCRIPTION:
Although acupuncture has been used in China and Japan for over 2000 years, it has only become increasingly important in Western medicine in the last few decades. A special form of acupuncture is "Yamamoto's New Skull Acupuncture" (YNSA), which was developed by Toshikatsu Yamamoto. Here, the needling is limited to the skull.

Acupuncture is a safe and almost painless procedure that is usually well tolerated. One indication might be the therapy of neurological diseases. Schockert and colleagues examined the effectiveness of YNSA in a placebo-controlled study. To investigate the effectiveness of cranial acupuncture, three fMRI sequences were performed: 1) without acupuncture, 2) sham acupuncture (acupressure without needling) and 3) YNSA acupuncture. The subjects (17 stroke patients with right hemisphere lesions and 19 healthy controls) were instructed to alternately make a fist (3s) and close it again (2s). There were a total of five blocks, each with a duration of 120s. Compared to sham acupuncture, cortical activations in motor, premotor and supplementary motor areas were observed during YNSA acupuncture.

In contrast to Schockert and colleagues, the planned study uses resting-state fMRI to determine whether YNSA acupuncture is associated with changes of functional connectivity within different resting-state networks.

ELIGIBILITY:
Inclusion Criteria:

* adults aged 18 to 65

Exclusion Criteria:

* mental disorders (dementia, depression)
* MRI contraindications
* claustrophobia
* weight > 120 kg

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers of both sexes aged 18-65 years
Sampling Method: Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2020-08-24 (Actual); Study Completion 2020-08-24 (Actual)

PRIMARY OUTCOMES:
Changed functional connectivity | 35 minutes
  Functional connectivity is measured using resting-state fMRI.

CONTACTS AND LOCATIONS:
Overall Officials: Jens D Rollnik, MD, Study Director — BDH-Clinic Hessisch Oldendorf
Locations (1):
- BDH-Clinic Hessisch Oldendorf, Hessisch Oldendorf, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Schockert T, Schnitker R, Boroojerdi B, Smith IQ, Yamamoto T, Vietzke K, Kastrau F. Cortical activation by Yamamoto new scalp acupuncture in the treatment of patients with a stroke: a sham-controlled study using functional MRI. Acupunct Med. 2010 Dec;28(4):212-4. doi: 10.1136/aim.2010.002683. Epub 2010 Oct 5. No abstract available. PMID 20923941